CLINICAL TRIAL: NCT04765384
Title: An Open-label, Phase 2 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Ad26.COV2.S in Healthy Pregnant Participants
Brief Title: A Study of Ad26.COV2.S in Healthy Pregnant Participants (COVID-19)
Acronym: HORIZON 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR108962; VAC31518COV2004 (Other: Janssen Research & Development, LLC); 2020-005330-14 (EudraCT Number)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Prevention
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Groups 1-4: Ad26.COV2.S (One Dose) (Experimental): Participants who are previously vaccinated (Group 1-3) and participants who are vaccine naïve (Group 4) will receive single dose of Ad26.COV2.S vaccine at standard dose level on Day 1. Participants from group 4 who are no longer pregnant may receive single booster dose of Ad26.COV2.S vaccine at standard dose level.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Participants will receive intramuscular (IM) injection of Ad26.COV2.S.
  Other Names: JNJ-78436735, Ad26COVS1

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of Ad26.COV2.S administered intramuscularly (IM) as a 1-dose schedule at the standard dose level in adult participants during the second and/or third trimester of pregnancy and (potentially) post-partum; to assess the humoral immune response in peripheral blood of adult participants to Ad26.COV2.S administered IM as a 1-dose schedule during the second and/or third trimester of pregnancy, 28 days after vaccination.

DETAILED DESCRIPTION:
There is an increased risk of severe coronavirus disease-2019 (COVID-19) during pregnancy, as well as an increased risk of adverse birth outcomes. Therefore, the aim of this study is to assess the safety, reactogenicity and immunogenicity of Ad26.COV2.S in adult participants in the second and/or third trimester of pregnancy. Ad26.COV2.S (also known as Ad26COVS1) is a monovalent vaccine composed of a recombinant, replication incompetent adenovirus type 26 (Ad26) vector, constructed to encode the S protein derived from a severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) clinical isolate, stabilized in its prefusion conformation. For each adult participant, the total study duration from screening until the last follow-up visit will be approximately 16 months. The study will consist of a screening phase (28 days), vaccination period (study period from vaccination to pregnancy completion/termination) and a follow-up period (up to 12 months post pregnancy completion/termination). For neonates/infants born to the participants in the study will be followed for approximately 12 months postpartum. Safety assessments will include immunogenicity assessments, physical examination, vital signs, clinical safety laboratory assessments, medical, obstetric and delivery history, pregnancy outcome, neonate safety assessment, adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI).

ELIGIBILITY:
Inclusion Criteria:

* If on medication for a condition, the medication dose must have been stable for at least 4 weeks preceding vaccination
* Participant must be healthy as confirmed by medical history, physical examination, vital signs, and obstetric history performed at Screening. Participant may have underlying illnesses, as long as the symptoms and signs are medically controlled
* Participant will be at second or third trimester of pregnancy, that is, Week 16 to Week 38 of gestation (inclusive), at the time of vaccination, based on ultrasound at the time of screening (or not longer than 10 days prior to vaccination if performed elsewhere)
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Participant either received their last COVID-19 vaccination with an authorized/licensed COVID-19 vaccine (at least 4 months prior to first study vaccination) or is COVID 19 vaccine-naïve

Exclusion Criteria:

* Participants with medical or obstetric histories that put them at higher risk for maternal or fetal complications (example, chronic pregnancy-related disorders, birth defects or genetic conditions during previous pregnancy)
* Participant with abnormal pregnancy screening test (example, ultrasound fetal abnormalities, maternal blood screen)
* Participant has a history of malignancy within 2 years before screening (exceptions are squamous, basal cell carcinomas of the skin, carcinoma in situ of the cervix, or malignancy, considered cured with minimal risk of recurrence)
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Participant has a history of any serious, chronic, or progressive neurological disorders or seizures including Guillain-Barre syndrome, with the exception of febrile seizures during childhood
* Participant has a positive diagnostic test result (polymerase chain reaction [PCR] based viral ribonucleic acid [RNA] detection) severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection at screening or Day 1 (if more than 4 days in between)
* Participant has a history of thrombosis with thrombocytopenia syndrome (TTS), including cerebral venous sinus thrombosis (CVST), or heparin-induced thrombocytopenia (HIT)
* Participant has a history of capillary leak syndrome (CLS)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (18):
- United States (4):
  - Medpharmics, LLC, Gulfport, Mississippi
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Medpharmics, LLC, Albuquerque, New Mexico
  - Maximos OB/GYN, League City, Texas
- Brazil (10):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Associacaode Ensino de Marilia LTDA - UNIMAR - Universidade de Marilia, Marília
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CEPCLIN, Natal
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Clinical Research College, São Paulo
  - CMPC - Consultoria Médica e Pesquisa Clínica, Sorocaba
- South Africa (4):
  - Ndlovu Elandsdoorn Site, Dennilton
  - Shandukani Research Centre, Johannesburg
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Soweto

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per plan, only adults were considered enrolled in the study.
Pre-assignment Details: Per change in planned analyses, combined analysis was performed for Groups 2 and 3 in both adults and neonates in order to protect and maintain the privacy/confidentiality of the single participant enrolled in Group 2. Each adult participant in Group 4 received booster dose at a different timepoint, that is, any day from Day 84 up to Day 364.
Groups:
- Group 1 (Adults): Ad26.COV2.S 5*10^10 vp: Adult participants from 2nd or 3rd trimester of pregnancy (Week 16 to Week 38 of gestation, inclusive), previously vaccinated (at least 4 months prior to receiving the study vaccine) exclusively with messenger Ribonucleic acid (mRNA) coronavirus disease 2019 (COVID-19) vaccine (primary vaccination [2-doses] or homologous booster vaccination) with COVID-19 mRNA vaccine (Pfizer-BioNTech or Moderna) received a single dose of the adenovirus type 26 (Ad26) vector, encoded with spike (S) protein from severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) (Ad26.COV2.S) 5*10^10 viral particles (vp) as intramuscular (IM) injection on Day 1.
- Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp: Adult participants from 2nd or 3rd trimester of pregnancy (Week 16 to Week 38 of gestation, inclusive), previously vaccinated (at least 4 months prior to receiving the study vaccine) with any regimen not included in Group 1 (non-mRNA or heterologous regimen) received a single dose of Ad26.COV2.S 5*10^10 vp as IM injection on Day 1.
- Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp: Adult participants from 2nd or 3rd trimester of pregnancy (Week 16 to Week 38 of gestation, inclusive), with no prior COVID-19 vaccination (vaccine- naive) received a single dose of Ad26.COV2.S 5*10^10 vp as IM injection on Day 1 followed by an optional single booster dose of Ad26.COV2.S 5*10^10 vp as IM injection on Booster Day 1 (any day between Day 84 and Day 364).
- Group 1 (Neonates and Infants): Neonates and infants of mothers from Group 1 (Adults) were followed up for up to 12 months postpartum. Neonates and infants in this group did not receive any active vaccination with Ad26.COV2.S 5*10^10 vp.
- Groups 2 and 3 (Neonates and Infants): Neonates and infants of mothers from Groups 2 and 3 (Adults) were followed up for up to 12 months postpartum. Neonates and infants in this group did not receive any active vaccination with Ad26.COV2.S 5*10^10 vp.
- Group 4 (Neonates and Infants): Neonates and infants of mothers from Group 4 (Adults) were followed up for up to 12 months postpartum. Neonates and infants in this group did not receive any active vaccination with Ad26.COV2.S 5*10^10 vp.
Period: Post-baseline: Adults
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp | Group 1 (Neonates and Infants) | Groups 2 and 3 (Neonates and Infants) | Group 4 (Neonates and Infants)
Started | 12 | 10 | 29 | 0 | 0 | 0
Adult Participants Who Received Booster Vaccination | 0 | 0 | 13 | 0 | 0 | 0
Group 2 | 0 | 1 | 0 | 0 | 0 | 0
Group 3 | 0 | 9 | 0 | 0 | 0 | 0
Completed | 10 | 8 | 23 | 0 | 0 | 0
Not Completed | 2 | 2 | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0 | 0 | 0
Period: Post-natal: Neonates and Infants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp | Group 1 (Neonates and Infants) | Groups 2 and 3 (Neonates and Infants) | Group 4 (Neonates and Infants)
Started | 0 | 0 | 0 | 10 | 8 | 29
Group 2 | 0 | 0 | 0 | 0 | 1 | 0
Group 3 | 0 | 0 | 0 | 0 | 7 | 0
Completed | 0 | 0 | 0 | 9 | 8 | 21
Not Completed | 0 | 0 | 0 | 1 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Parent Or Guardian | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Per planned analysis, data for baseline characteristics were collected and analyzed for the full analysis set - adults (FAS-A) which included all enrolled adult participants with at least one vaccine administration documented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp | Total
Number analyzed (Participants) | 12 | 10 | 29 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.42) | 24.2 (3.61) | 25.4 (5.29) | 24.9 (4.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 29 | 51
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 10 | 26
  Not Hispanic or Latino | 2 | 4 | 18 | 24
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 9 | 16
  White | 8 | 3 | 18 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 12 | 9 | 11 | 32
  South Africa | 0 | 1 | 4 | 5
  United States | 0 | 0 | 14 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Adult Participants With Solicited Local Adverse Events (AEs) for 7 Days Post First Vaccination
Description: Number of adult participants with solicited local AEs for 7 days post first vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were pre-defined as local (at the injection site) AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post first vaccination (day of first vaccination and the subsequent 7 days). Solicited local AEs are injection site pain/tenderness, erythema, swelling at the vaccination site.
Time Frame: From first vaccination on Day 1 up to 7 days post first vaccination (up to Day 8)
Population: Full Analysis Set - Adults (FAS-A) included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 10 | 5 | 20

2. Primary Outcome: Number of Adult Participants With Solicited Systemic AEs for 7 Days Post First Vaccination
Description: Number of adult participants with solicited systemic AEs for 7 days post first vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were predefined as systemic AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post first vaccination. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post first vaccination (day of first vaccination and the subsequent 7 days) for the following solicited systemic AEs: fatigue, headache, nausea, myalgia.
Time Frame: From first vaccination on Day 1 up to 7 days post first vaccination (up to Day 8)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 10 | 4 | 20

3. Primary Outcome: Number of Adult Participants With Unsolicited AEs for 28 Days Post First Vaccination
Description: Number of adult participants with unsolicited AEs for 28 days post first vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were defined as AEs for which the participants were not specifically questioned in the participant's reactogenicity diary.
Time Frame: From first vaccination on Day 1 up to 28 days post first vaccination (up to Day 29)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 7 | 4 | 10

4. Primary Outcome: Number of Adult Participants With Serious Adverse Events (SAEs) From First Vaccination Until End of the Study (EOS)
Description: Number of adult participants with SAEs from first vaccination until EOS were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAEs were defined as any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From first vaccination on Day 1 until end of study (up to post-partum [PP] Day 366 [Day 15 up to Day 554])
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 4 | 2 | 3

5. Primary Outcome: Number of Adult Participants With Adverse Events of Special Interest (AESIs) From First Vaccination Until EOS
Description: Number of adult participants with AESIs from first vaccination until EOS were reported. Thrombosis with thrombocytopenia syndrome (TTS) in adults was considered an AESI in this study. TTS is a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia.
Time Frame: From first vaccination on Day 1 until end of study (up to PP Day 366 [Day 15 up to Day 554])
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 0 | 0 | 0

6. Primary Outcome: Number of Adult Participants With Medically Attended Adverse Events (MAAEs) Until 6 Months Post First Vaccination
Description: Number of adult participants with MAAEs until 6 months post first vaccination was reported. MAAEs were defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically attended visits. New onset of chronic diseases was collected as part of the MAAEs.
Time Frame: From first vaccination on Day 1 until 6 months post first vaccination (up to Day 183)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 6 | 2 | 7

7. Primary Outcome: Number of Adult Participants With AEs Leading to Study Discontinuation
Description: Number of adult participants with AEs leading to study discontinuation were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. All AEs leading to discontinuation from the study (regardless of the causal relationship) were reported for all adult participants from the moment of first vaccination until completion of the participant's last study-related procedure.
Time Frame: From first vaccination on Day 1 until end of study (up to PP Day 366 [Day 15 up to Day 554])
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants | 0 | 0 | 0

8. Primary Outcome: Serological Response to Vaccination as Measured by S-Enzyme-linked Immunosorbent Assay (S-ELISA) in Adult Participants 28 Days Post First Vaccination
Description: Serological response to vaccination as measured by S-ELISA in adult participants 28 days post first vaccination was reported.
Time Frame: 28 days post first vaccination on Day 1 (at Day 29)
Population: Per-protocol Immunogenicity-Adults (PPI-A) set included all vaccinated adult participants for whom immunogenicity data were available excluding adult participants with major protocol deviations that were expected to impact the immunogenicity outcomes. Here, "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 9 | 8 | 24
ELISA units per milliliter (EU/mL) | 19179 [10137 to 36284] | 12335 [8796 to 17299] | 5906 [2784 to 12529]

9. Secondary Outcome: Group 4: Number of Adult Participants With Solicited Local AEs for 7 Days Post Booster Vaccination
Description: Number of adult participants with solicited local AEs for 7 days post booster vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were pre-defined as local (at the injection site) AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post booster vaccination (day of booster vaccination and the subsequent 7 days). Solicited local AEs are: injection site pain/tenderness, erythema, swelling at the vaccination site.
Time Frame: 7 days post booster vaccination (Day 84 up to Day 371)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented. Data for this outcome measure was planned to be collected and analyzed only for the participants in arm "Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp", as only this arm received the booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 6

10. Secondary Outcome: Group 4: Number of Adult Participants With Solicited Systemic AEs for 7 Days Post Booster Vaccination
Description: Number of adult participants with solicited systemic AEs for 7 days post booster vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were predefined as systemic AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post booster vaccination. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (day of booster vaccination and the subsequent 7 days) for the following solicited systemic AEs: fatigue, headache, nausea, myalgia.
Time Frame: 7 days post booster vaccination (Day 84 up to Day 371)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 7

11. Secondary Outcome: Group 4: Number of Adult Participants With Unsolicited AEs for 28 Days Post Booster Vaccination
Description: Number of adult participants with unsolicited AEs for 28 days post booster vaccination was reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were defined as AEs for which the participants were not specifically questioned in the participant's reactogenicity diary.
Time Frame: 28 days post booster vaccination (Day 84 up to Day 392)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 2

12. Secondary Outcome: Group 4: Number of Adult Participants With SAEs Post Booster Vaccination Until EOS
Description: Number of adult participants with SAEs post booster vaccination until EOS were reported. AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAE were defined as any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From booster vaccination (Day 84 up to Day 364) until EOS (up to PP Day 366 [Day 366 up to Day 554])
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 0

13. Secondary Outcome: Group 4: Number of Adult Participants With AESIs Post Booster Vaccination Until EOS
Description: Number of adult participants with AESI post booster vaccination until EOS were reported. Thrombosis with thrombocytopenia syndrome (TTS) in adults was considered an AESI in this study. TTS is a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia.
Time Frame: From booster vaccination (Day 84 up to Day 364) until EOS (up to PP Day 366 [Day 366 up to Day 554])
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 0

14. Secondary Outcome: Group 4: Number of Adult Participants With MAAEs Until 6 Months Post Booster Vaccination
Description: Number of adult participants with MAAEs until 6 months post booster vaccination were reported. MAAEs were defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically attended visits. New onset of chronic diseases was collected as part of the MAAEs.
Time Frame: 6 months post booster vaccination (Day 84 up to Day 546)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 0

15. Secondary Outcome: Group 4: Number of Adult Participants With AEs Leading to Study Discontinuation Post Booster Vaccination Until EOS
Description: Number of adult participants with AEs leading to study discontinuation post booster vaccination until EOS were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. All AEs leading to discontinuation from the study (regardless of the causal relationship) were reported for all adult participants from the moment of booster vaccination until completion of the participant's last study-related procedure.
Time Frame: From post booster vaccination (Day 84 up to Day 364) until EOS (up to PP Day 366 [Day 366 up to Day 554])
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
Participants | 0

16. Secondary Outcome: Number of Adult Participants With Pregnancy Outcomes
Description: Number of adult participants with pregnancy outcomes were reported. Pregnancy outcomes in adult participants included live term birth, live preterm birth, stillbirth, and abortion.
Time Frame: From first vaccination on Day 1 until PP Day 1 (Day 7 up to Day 163)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 10 | 8 | 29
Participants
  Live Term Birth | 10 | 7 | 26
  Live Preterm Birth | 0 | 1 | 3
  Stillbirth | 0 | 0 | 0
  Abortion | 0 | 0 | 0

17. Secondary Outcome: Number of Adult Participants With Pregnancy Related AEs Throughout Pregnancy
Description: Number of adult participants with pregnancy related AEs throughout pregnancy were reported. Pregnancy related AEs in adult participants were collected based on 2 baseline gestational age groups (adult participants who received vaccination at 16 to 27 weeks [>=16 weeks to <28 weeks] and at 28 to 38 weeks [>=28 weeks to <=38 weeks]) and included gestational hypertension, foetal growth restriction, haemorrhage in pregnancy, polyhydramnios, pre-eclampsia, premature rupture of membranes, preterm premature rupture of membranes, bradycardia foetal, premature baby, amniorrhexis, foetalgrowth restriction, amniotic fluid volume decreased.
Time Frame: From first vaccination on Day 1 until PP Day 1 (Day 7 up to Day 163)
Population: FAS-A included all enrolled adult participants with at least one vaccine administration documented. Here "n"(number analyzed) signifies number of participants analyzed for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 12 | 10 | 29
Participants
  Gestational Age: 16-27 weeks: number analyzed (Participants) | 8 | 5 | 14
  Gestational Age: 16-27 weeks | 4 | 2 | 3
  Gestational Age: 28-38 weeks: number analyzed (Participants) | 4 | 5 | 15
  Gestational Age: 28-38 weeks | 1 | 3 | 1

18. Secondary Outcome: Serological Response to First Vaccination as Measured by S-ELISA in Adult Participants at All Blood Collection Timepoints Post First Vaccination
Description: Serological response to first vaccination as measured by S-ELISA at all blood collection timepoints post first vaccination were reported.
Time Frame: Day 1, Day 29, PP Day 1 (Day 7 up to Day 163), PP Day 183 (Day 189 up to Day 345)
Population: PPI-A set included all vaccinated adult participants for whom immunogenicity data were available excluding adult participants with major protocol deviations that were expected to impact the immunogenicity outcomes. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n" (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 9 | 9 | 29
ELISA Units per milliliter (EU/mL)
  Day 1 | 10977 [7375 to 16336] | 2927 [1266 to 6770] | 197 [101 to 383]
  Day 29: number analyzed (Participants) | 9 | 8 | 24
  Day 29 | 19179 [10137 to 36284] | 12335 [8796 to 17299] | 5906 [2784 to 12529]
  PP Day 1 (Day 7 up to Day 163): number analyzed (Participants) | 6 | 7 | 27
  PP Day 1 (Day 7 up to Day 163) | 16733 [8776 to 31903] | 10179 [5418 to 19123] | 4025 [2115 to 7659]
  PP Day 183 (Day 189 up to Day 345): number analyzed (Participants) | 8 | 7 | 23
  PP Day 183 (Day 189 up to Day 345) | 12704 [8852 to 18233] | 8846 [5851 to 13373] | 4698 [2652 to 8324]

19. Secondary Outcome: Serological Response to First Vaccination as Measured by Virus Neutralization Assay (VNA) Titers, 28 Days in Adult Participants Post First Vaccination
Description: Serological response to first vaccination measured by VNA titers at 28 days in adult participants post first vaccination was reported. Data were expressed as 50 percent (%) inhibitory concentration (IC50) units.
Time Frame: 28 days post first vaccination on Day 1 (at Day 29)
Population: PPI-A set included all vaccinated adult participants for whom immunogenicity data were available excluding adult participants with major protocol deviations that were expected to impact the immunogenicity outcomes. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 9 | 8 | 24
titers | 7233 [3410 to 15342] | 5527 [3106 to 9834] | 1601 [639 to 4012]

20. Secondary Outcome: Group 4: Serological Response to Booster Vaccination Measured by Binding (S-ELISA) Antibody Titers in Adult Participants at Blood Collection Time Points Post Booster Vaccination
Description: Serological response to vaccination as measured by binding (S-ELISA) antibody titers in adult participants at blood collection time points post booster vaccination were reported.
Time Frame: Booster Day 1 (Day 84 up to Day 364), Booster Day 29 (Day 112 up to Day 392)
Population: PPI-A set included all vaccinated adult participants with available immunogenicity data excluding participants with major protocol deviations that impact immunogenicity outcomes. Data for this outcome measure was planned to be collected and analyzed only for the participants in arm "Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp", as only this arm received the booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
ELISA Units per milliliter (EU/mL)
  Booster Day 1 (Day 84 up to Day 364) | 4204 [1996 to 8857]
  Booster Day 29 (Day 112 up to Day 392) | 7213 [4417 to 11780]

21. Secondary Outcome: Group 4: Serological Response to Booster Vaccination Measured by Neutralizing (VNA) Antibody Titers in Adult Participants at Blood Collection Time Points Post Booster Vaccination
Description: Serological response to booster vaccination measured by neutralizing VNA antibody titers in adult participants at blood collection time points post booster vaccination were reported. Data were expressed as IC50 units.
Time Frame: Booster Day 1 (Day 84 up to Day 364), Booster Day 29 (Day 112 up to Day 392)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp
Number analyzed (Participants) | 13
titers
  Booster Day 1 (Day 84 up to Day 364): number analyzed (Participants) | 12
  Booster Day 1 (Day 84 up to Day 364) | 1299 [419 to 4029]
  Booster Day 29 (Day 112 up to Day 392) | 3203 [1166 to 8802]

22. Secondary Outcome: Serological Response to Vaccination as Measured by S-ELISA at Birth (That is, in Cord Blood) and at 2 Months and 6 Months of Age in Neonates and Infants Born to Adult Participants
Description: Serological response to vaccination as measured by S-ELISA at birth (that is, in cord blood) and at 2 months and 6 months of age in neonates and infants born to adult participants were reported.
Time Frame: At birth (postnatal [PN] Day 1 [Day 7 up to Day 163]), 2 months (up to PN Day 61 [Day 67 up to Day 223]) and 6 months (up to PN Day 183 [Day 189 up to Day 345])
Population: Per-protocol immunogenicity- non-vaccinated neonates/infants (PPI-NVN) included all non-vaccinated neonates/infants born to Ad26.COV2.S vaccinated adult participants for whom immunogenicity data were available. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Groups:
- Group 1 (Neonates and Infants): Mother's With Prior mRNA: Neonates and infants of mothers with prior mRNA COVID-19 vaccination. Participants received no active vaccination with Ad26.COV2.S 5*10^10 vp in this study. Neonates/infants born to the participants previously vaccinated with mRNA COVID-19 vaccine (primary vaccination [2-doses] or homologous booster vaccination) were followed for approximately 12 months postpartum.
- Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination: Neonates and infants of mothers with prior mRNA COVID-19 vaccination. Participants received no active vaccination with Ad26.COV2.S 5*10^10 vp in this study. Neonates/infants born to the participants a primary vaccination (1-dose) or homologous booster vaccination and COVID-19 vaccination irrespective of previous schedule and vaccine (included heterologous regimens) and excluded schedules for Groups 1 and 2 were followed for 12 months postpartum.
- Group 4 (Neonates and Infants) of Vaccine-naive Mother's: Neonates and infants of mother's who were vaccine-naive received no active vaccination with Ad26.COV2.S 5*10^10 vp in this study. Neonates/infants born to the participants previously not vaccinated with COVID-19 vaccine were followed for 12 months postpartum.
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 7 | 6 | 23
ELISA Units per milliliter (EU/mL)
  PN Day 1 [Day 7 up to Day 163]): number analyzed (Participants) | 6 | 6 | 23
  PN Day 1 [Day 7 up to Day 163]) | 17327 [9676 to 31027] | 11540 [6862 to 19406] | 4013 [1758 to 9162]
  PN Day 61 [Day 67 up to Day 223]): number analyzed (Participants) | 7 | 5 | 23
  PN Day 61 [Day 67 up to Day 223]) | 4021 [1856 to 8711] | 3520 [1740 to 7123] | 2996 [1697 to 5289]
  PN Day 183 [Day 189 up to Day 345): number analyzed (Participants) | 6 | 6 | 22
  PN Day 183 [Day 189 up to Day 345) | 529 [230 to 1216] | 477 [217 to 1048] | 795 [390 to 1618]

23. Secondary Outcome: Serological Response to Vaccination as Measured by VNA Titers at Birth (That is, in Cord Blood) in Neonates and Infants Born to Adult Participants
Description: Serological response to vaccination as measured by VNA titers at birth (that is, in cord blood) in neonates and infants born to adult participants were reported. Data were expressed as IC50 units.
Time Frame: At Birth (PN Day 1 [Day 7 up to Day 163])
Population: Per-protocol immunogenicity- non-vaccinated neonates/infants (PPI-NVN) included all non-vaccinated neonates/infants born to Ad26.COV2.S vaccinated adult participants for whom immunogenicity data were available. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 6 | 6 | 26
titers | 3788 [1776 to 8082] | 3756 [1740 to 8106] | 658 [236 to 1834]

24. Secondary Outcome: Number of Neonates and Infants With SAEs (Including MIS-C) From Birth Up to 12 Months of Age in Neonates and Infants Born to Adult Participants
Description: An AE is any untoward medical occurrence in participants in the study that does not necessarily have a causal relationship with pharmaceutical/biological agent under study. SAE: any untoward medical occurrence that resulted in following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important. MIS-C: a serious and potentially fatal condition in infants and children with SARS-CoV-2, which resulted in inflammation involving multiple organs. Symptoms of MIS-C: persistent fever, fatigue and signs and symptoms including multiorgan systems (cardiac, gastrointestinal, renal, hematologic, dermatologic, neurologic) involvement, elevated inflammatory markers and, in severe cases, hypotension and shock.
Time Frame: From birth (PN Day 1 [Day 7 up to Day 163]) up to 12 months of age (up to PN Day 366 [Day 372 up to Day 528])
Population: Full Analysis Set - Non-vaccinated Neonates/Infants (FAS-NVN) included all non-vaccinated neonates/infants born to Ad26.COV2.S vaccinated adult participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 10 | 8 | 29
Participants | 3 | 4 | 4

25. Secondary Outcome: Number of Neonates and Infants With AESIs From Birth Until 12 Months of Age in Neonates and Infants Born to Adult Participants
Description: Number of neonates and infants with AESIs from birth until 12 months of age in neonates and infants born to adult participants were reported. TTS is a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia.
Time Frame: From birth (PN Day 1 [Day 7 up to Day 163]) until 12 months of age (up to PN Day 366 [Day 372 up to Day 528])
Population: FAS-NVN included all non-vaccinated neonates/infants (NVN) born to Ad26.COV2.S vaccinated adult participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 10 | 8 | 29
Participants | 0 | 0 | 0

26. Secondary Outcome: Number of Neonates and Infants With MAAEs From Birth Until 6 Months of Age in Neonates and Infants Born to Adult Participants
Description: Number of neonates and infants with MAAEs from birth until 6 months of age in neonates and infants born to adult participants were reported. MAAEs were defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically attended visits. New onset of chronic diseases were collected as part of the MAAEs.
Time Frame: From birth (PN Day 1 [Day 7 up to Day 163]) until 6 months of age (up to PN 183 [Day 189 up to Day 345])
Population: FAS-NVN included all non-vaccinated neonates/infants (NVN) born to Ad26.COV2.S vaccinated adult participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 10 | 8 | 29
Participants | 5 | 4 | 5

27. Secondary Outcome: Number of Neonates and Infants With AEs Leading to Study Discontinuation From Birth Until Study Discontinuation
Description: Number of neonates and infants with AEs leading to study discontinuation from birth until study discontinuation were reported. An AE is any untoward medical occurrence in participants who does not necessarily have a causal relationship with pharmaceutical/biological agent under study. All AEs leading to discontinuation from the study (regardless of the causal relationship) were reported for all neonates and infants.
Time Frame: From birth (PN Day 1 [Day 7 up to Day 163]) until study discontinuation (until 12 months of age [up to PN Day 366 {Day 372 up to Day 528}])
Population: FAS-NVN included all non-vaccinated neonates/infants (NVN) born to Ad26.COV2.S vaccinated adult participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 10 | 8 | 29
Participants | 0 | 0 | 0

28. Secondary Outcome: Number of Neonates and Infants With Different Birth Outcomes From Birth Up to 12 Months of Age
Description: Number of neonates and infants with different birth outcomes from birth until 12 months of age were reported. Neonate/infant outcomes included normal neonate, term neonate with (or without) complications, preterm neonate with (or without) complications, neonatal infection, respiratory distress, congenital anomalies, neonatal death, low birth weight, and small for gestational age.
Time Frame: From birth (PN Day 1 [Day 7 up to Day 163]) up to 12 months of age (up to PN Day 366 [Day 372 up to Day 528])
Population: FAS-NVN included all non-vaccinated neonates/infants (NVN) born to Ad26.COV2.S vaccinated adult participants. Here 'N' (Number of participants analyzed) signifies the number of participants who completed the neonatal medical history form and were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): Mother's With Prior mRNA | Group 2 & 3 (Neonates and Infants): Mother's With Prior Other COVID-19 Vaccination | Group 4 (Neonates and Infants) of Vaccine-naive Mother's
Number analyzed (Participants) | 10 | 8 | 29
Participants
  Normal neonate: number analyzed (Participants) | 10 | 7 | 29
  Normal neonate | 9 | 7 | 25
  Term neonate with complications: number analyzed (Participants) | 10 | 7 | 29
  Term neonate with complications | 0 | 0 | 1
  Preterm neonate with complications: number analyzed (Participants) | 10 | 7 | 29
  Preterm neonate with complications | 0 | 0 | 1
  Neonatal infection: number analyzed (Participants) | 10 | 7 | 29
  Neonatal infection | 0 | 0 | 0
  Respiratory distress: number analyzed (Participants) | 10 | 7 | 29
  Respiratory distress | 0 | 0 | 0
  Congenital anomalies: number analyzed (Participants) | 10 | 7 | 29
  Congenital anomalies | 0 | 0 | 0
  Neonatal death: number analyzed (Participants) | 10 | 7 | 29
  Neonatal death | 0 | 0 | 0
  Low birth weight: number analyzed (Participants) | 10 | 7 | 29
  Low birth weight | 1 | 0 | 0
  Small for gestational age: number analyzed (Participants) | 10 | 7 | 29
  Small for gestational age | 0 | 0 | 0
  Preterm neonate without complications: number analyzed (Participants) | 10 | 7 | 29
  Preterm neonate without complications | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adult participants: From first vaccination on Day 1 until EOS (up to PP Day 366 [Day 15 up to Day 554]), Neonates & Infants: From birth (PN Day 1 [Day 7 up to Day 163]) up to 12 months of age (up to PN Day 366 [Day 372 up to Day 528]), Solicited AEs: From first vaccination on Day 1 until 7 days post first vaccination (up to Day 8), Group 4: Solicited AEs (booster vaccination): 7 days post booster vaccination (Day 84 up to Day 371)
Description: Adult participants: FAS-A included all enrolled adult participants with at least one vaccine administration documented.
  Neonates and Infants: FAS-NVN included all non-vaccinated neonates/infants born to Ad26.COV2.S vaccinated adult participants.
  For solicited AEs, participants at risk=0 (neonates and infants) signifies that no solicited AEs were collected for infants and neonates since they didn't receive any study vaccination during the study.
Arm/Group | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp | Group 1 (Neonates and Infants) | Groups 2 and 3 (Neonates and Infants) | Group 4 (Neonates and Infants)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/29 | 1/10 | 0/8 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/12 | 2/10 | 3/29 | 3/10 | 4/8 | 4/29
Other Adverse Events (participants affected / at risk) | 12/12 | 8/10 | 27/29 | 7/10 | 5/8 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp (N=12) | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp (N=10) | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp (N=29) | Group 1 (Neonates and Infants) (N=10) | Groups 2 and 3 (Neonates and Infants) (N=8) | Group 4 (Neonates and Infants) (N=29)
Bradycardia Foetal (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholestasis of Pregnancy (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neonatal Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arboviral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhage in Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Placental Insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Preterm Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Perinatal Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient Tachypnoea of the Newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 (Adults): Ad26.COV2.S 5*10^10 vp (N=12) | Groups 2 and 3 (Adults): Ad26.COV2.S 5*10^10 vp (N=10) | Group 4 (Adults): Vaccine-naive: Ad26.COV2.S 5*10^10 vp (N=29) | Group 1 (Neonates and Infants) (N=10) | Groups 2 and 3 (Neonates and Infants) (N=8) | Group 4 (Neonates and Infants) (N=29)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Solicited) (Gastrointestinal disorders) | 5 | 1 | 11 | 0/0 | 0/0 | 0/0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 2
Chills (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 0 | 0 | 1
Fatigue (Solicited) (General disorders) | 9 | 2 | 19 | 0/0 | 0/0 | 0/0
Malaise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (Solicited) (General disorders) | 0 | 1 | 2 | 0/0 | 0/0 | 0/0
Vaccination Site Erythema (Solicited) (General disorders) | 3 | 0 | 1 | 0/0 | 0/0 | 0/0
Vaccination Site Pain (Solicited) (General disorders) | 10 | 5 | 20 | 0/0 | 0/0 | 0/0
Vaccination Site Swelling (Solicited) (General disorders) | 2 | 0 | 2 | 0/0 | 0/0 | 0/0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Neonatal Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 1 | 3 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 0 | 2 | 4 | 1 | 6
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Toxoplasmosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Amniotic Fluid Volume Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood Sodium Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Coombs Indirect Test Positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Mns System Antibodies Positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 7 | 1 | 14 | 0/0 | 0/0 | 0/0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0
Headache (Solicited) (Nervous system disorders) | 8 | 4 | 17 | 0/0 | 0/0 | 0/0
Foetal Growth Restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1 | 5
Placental Insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Retained Placenta or Membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Uterine Contractions During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Uterine Hypotonus (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0 | 0
Perinatal Depression (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Sample size for safety and immunogenicity analyses was low. In addition, further subdivision into subgroups by baseline serostatus and by baseline gestational age led to a further decrease in vaccination group sizes, making it difficult to draw any meaningful conclusions for the subgroup analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04765384/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04765384/SAP_001.pdf